CLINICAL TRIAL: NCT05407584
Title: Oregovomab and Non-platinum Chemotherapy in PARP Inhibitor Resistant Ovarian, Fallopian Tube, or Primary Peritoneal Cancer Patients Not Candidate for Platinum Retreatment: a Multicenter, Two-cohort, Single-arm Phase 2 Trial
Brief Title: Oregovomab and PLD in PARP Inhibitor Resistant Ovarian, Fallopian Tube, or Primary Peritoneal Cancer Patients Not Candidate for Platinum Retreatment
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Collaborators: CanariaBio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2022-0430
Record Dates: First submitted 2022-06-01; First posted 2022-06-07 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: PARP Inhibitor Resistant Ovarian, Fallopian Tube, or Primary Peritoneal Cancer Patients Not Candidate for Platinum Retreatment
Keywords: PARP inhibitor Resistant; platinum resistant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1(1-3 prior line of chemotherapy) (Experimental): Oregovomab and PLD is synergistic in PARPi-resistant recurrent ovarian cancer.
  Interventions: Drug: Orevogomab+PLD
- Cohort2 (>3prior line of chemotherapy) (Experimental): Oregovomab and Paclitaxel show synergistic in PARPi-resistant recurrent ovarian cancer.
  Interventions: Drug: Orevogomab+Paclitaxel

INTERVENTIONS:
Drug: Orevogomab+PLD — PLD (40 mg / m2 IV over three hours in one day) to be repeated till progression or unacceptable toxicity every four weeks (28 days)
  Investigational agent (Oregovomab): 2 mg diluted in 50 mL saline for injection administered IV following PLD over approximately 20 (acceptable range 15-30) minutes for a total of 5 scheduled injections, one each at Cycle 1, Cycle 2, Cycle 3, Cycle 5, and Cycle 7
  Arms: Cohort 1(1-3 prior line of chemotherapy)
Drug: Orevogomab+Paclitaxel — paclitaxel (80 mg / m2 IV over three hours in one day) to be repeated till progression or unacceptable toxicity every four weeks on day 1, 8, 15
  Investigational agent (Oregovomab): 2 mg diluted in 50 mL saline for injection administered IV following paclitaxel over approximately 20 (acceptable range 15-30) minutes for a total of 5 scheduled injections, one each at Cycle 1, Cycle 2, Cycle 3, Cycle 5, and Cycle 7
  Arms: Cohort2 (>3prior line of chemotherapy)

SUMMARY:
This study is phase II, open label, clinical trial to determine the efficacy of Oregovomab and non-platinum chemotherapy in PARP inhibitor resistant ovarian, fallopian tube, or primary peritoneal cancer patients who were not suitable for platinum retreatment.

Patients who have received one to three prior lines of chemotherapy are to be assigned to Cohort 1 (oregovamab 2 mg [C1,2,3,5,7 for five doses] + pegylated liposomal doxorubicin [PLD] 40 mg/m2 q4w, n=28), while patients who have received more than three prior lines of chemotherapy are to be assigned to Cohort 2 (oregovamab 2 mg [C1,2,3,5,7 for five doses] + weekly paclitaxel 80 mg/m2 [D1,8,15 q4w], n=28). A total of 56 patients will be recruited and treated with oregovomab + PLD / weekly paclitaxel until disease progression, unacceptable toxicity, or withdrawal of patient consent. The primary endpoint is objective response rate by RECIST 1.1.

DETAILED DESCRIPTION:
This study is a two-cohort, single arm phase II study in patients with PARP inhibitor-resistant ovarian, fallopian tube, or primary peritoneal cancer. The efficacy and safety of five administrations of Oregovomab 2mg IV in combination with non-platinum chemotherapy will be evaluated with recurrent ovarian cancer who have progressed with prior PARP inhibitor treatment.

Patients with disease under study will be screened for eligibility during the period 28 days immediately prior to starting study drug on Day 1. Laboratory and radiological assessments performed as part of standard of care before signing informed consent may be used if performed within the screening/baseline time window.

During this time, the inclusion and exclusion criteria will be assessed and all screening assessments, laboratory tests, and procedures will be performed.

Cohort 1(1-3 prior line of chemotherapy) PLD (40 mg / m2 IV over three hours in one day) to be repeated till progression or unacceptable toxicity every four weeks (28 days) Investigational agent (Oregovomab): 2 mg diluted in 50 mL saline for injection administered IV following PLD over approximately 20 (acceptable range 15-30) minutes for a total of 5 scheduled injections, one each at Cycle 1, Cycle 2, Cycle 3, Cycle 5, and Cycle 7

Cohort2 (>3prior line of chemotherapy) paclitaxel (80 mg / m2 IV over three hours in one day) to be repeated till progression or unacceptable toxicity every four weeks on day 1, 8, 15

Investigational agent (Oregovomab): 2 mg diluted in 50 mL saline for injection administered IV following paclitaxel over approximately 20 (acceptable range 15-30) minutes for a total of 5 scheduled injections, one each at Cycle 1, Cycle 2, Cycle 3, Cycle 5, and Cycle 7

ELIGIBILITY:
Inclusion Criteria:

1. Adults 20 years old or older.
2. Subjects with histologically confirmed epithelial adenocarcinoma of ovarian, fallopian tube or peritoneal origin.
3. Eligible histologic epithelial cell types: high grade serous adenocarcinoma, high grade endometrioid adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, , and low-grade adenocarcinoma, or adenocarcinoma not otherwise specified (N.O.S.).

   [only up to 5 patients with non-high grade serous carcinoma will be included]
4. Prior PARP inhibitor exposure (progressed through a prior PARP inhibitor)
5. CA-125 ≥ 50 U/ml
6. Prior platinum-based chemotherapy.
7. Cohort 1 : 1-3 prior lines of therapies / Cohort 2 : Previous treatments of the 4th line or more.
8. Not eligible for platinum re-treatment (prior allergic reaction or residual toxicity, patients who are not able to receive (in the physician's opinion) or willing to receive platinum treatment and platinum resistant patients)
9. Received prior bevacizumab or not eligible for bevacizumab due to medical.
10. Adequate bone marrow function:

    1. Absolute neutrophil count (ANC) ≥ 1,500/μL
    2. Platelets ≥ 100,000/μL
    3. Hemoglobin ≥ 8.0 g/dL (Note: Blood transfusion is permitted up to 48 hours before first dose of study treatment).
11. Adequate liver function:

    1. Bilirubin < 1.5 times upper limit normal (ULN)
    2. Lactate Dehydrogenase (LDH), SGOT/AST and SGPT/ALT < 2.5 times ULN
12. Adequate renal function:

    a. Creatinine ≤ 1.5 times ULN
13. ECOG Performance Status of 0 or 1.
14. For women of childbearing potential, must be willing to avoid pregnancy by using a highly effective method of contraception from the first dose of study treatment to 60 days after last dose of study treatment.
15. Sign informed consent and authorization permitting release of personal health information.

Exclusion Criteria:

1. Participant has mucinous, germ cell, or borderline tumor of the ovary.
2. Female subjects who are lactating and breastfeeding, or have a positive serum pregnancy test within 7 days prior to the first dose of study treatment.
3. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
4. Active autoimmune disease, such as rheumatoid arthritis, systemic lupus erythematosus (SLE), ulcerative colitis, Crohn's Disease, multiple sclerosis (MS), or ankylosing spondylitis requiring active disease modifying treatment.
5. Known allergy to murine proteins or hypersensitivity to any of the excipients of the oregovomab and PLD.
6. Chronically treated with immunosuppressive drugs such as cyclosporine, adrenocorticotropic hormone (ACTH), etc.
7. Chronic therapeutic corticosteroid use, defined as > 5 days of prednisone or equivalent, with the exception of inhalers or those on a pre-planned steroid taper.
8. Recognized acquired, hereditary, or congenital immunodeficiency disease, including cellular immunodeficiencies, hypogammaglobulinemia or dysgammaglobulinemia.
9. Clinically significant active infection(s) at the time of screening.
10. Any of the following conditions (on-study testing is not required):

    1. Known HIV-infected subjects unless on effective anti-retroviral therapy with an undetectable viral load within 6 months, or
    2. Known or suspected hepatitis B if active infection (patients with chronic hepatitis B infection must have an undetectable HBV viral load on suppressive therapy, if indicated; positive surface antibody alone is not an exclusion), or
    3. Known or suspected hepatitis C infection which has not been treated and cured unless currently on treatment with an undetectable viral load).
11. Uncontrolled or life-threatening diseases compromising safety evaluation.
12. Participant has a known additional malignancy that is progressing or has required active treatment within the past 2 years.

    Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ, endometrial carcinoma) that have undergone potentially curative therapy are not excluded.

    Note: Participants with synchronous primary endometrial cancer or a past history of primary endometrial cancer that met the following conditions are not excluded: Stage not greater than IA: no more than superficial myometrial invasion.
13. Contraindications to the use of pressor agents
14. History or evidence upon physical examination of CNS disease, seizures not controlled with standard medical therapy, or any brain metastases.
15. Any of the following cardiovascular conditions:

    1. Acute myocardial infarction within 6 months before the first dose of study treatment.
    2. Current history of New York Heart Association (NYHA) Class III or IV heart failure (see Appendix H).
    3. Evidence of current uncontrolled cardiovascular conditions including cardiac arrhythmias, angina, pulmonary hypertension, or electrocardiographic clinically significant findings.
16. Unable to read or understand or unable to sign the necessary written consent before starting treatment.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 56 (Estimated)
Dates: Start 2022-07-05 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Confirmed ORR | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  based on radiographically confirmed response according to CR+PR rate based on RECIST v1.1 as determined by the investigator

SECONDARY OUTCOMES:
progression-free survival | Up to 1 years
  PFS is calculated as the interval in months from the date of enrollment to the date of disease progression or the date of death, whichever comes first.
Overall survival (OS) | Up to 1 years
  Overall survival (OS) will be calculated using the date of death OS is calculated as the interval in months from the date of enrollment to the date of death.
Time to first Subsequent Therapy | The date of first documented first subsequent treatment or date of death, assessed up to 72 months
  TFST, defined as time from the date of enrollment into the study to second anti-cancer therapy start date following study treatment completion, treatment exit [EOT] or death, will be determined.
Time to Second Subsequent Therapy | The date of first documented second subsequent treatment assessed up to 72 months
  TSST, defined as time from the date of enrollment into the study to third anti-cancer therapy start date following study treatment completion, treatment exit [EOT] or death, will be determined.
Duration of response | Up to 1 years
  DOR, defined as the time from the first occurrence of a documented objective response to disease progression or death from any cause (whichever occurs first), as determined by the investigator according to RECIST v1.1
second objective disease progression | Up to 1 years
  PFS2, defined as the time from enrollment into the study to the earlier date of progression on next-line therapy or death from any cause, will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Yun Lee, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park J, Cho HW, Lim MC, Choi CH, Lee JY. OPERA: a phase II trial of oregovomab plus non-platinum chemotherapy in PARP inhibitor/platinum-resistant ovarian cancer. Future Oncol. 2024;20(26):1893-1899. doi: 10.1080/14796694.2024.2357533. Epub 2024 Jun 28. PMID 38940373